CLINICAL TRIAL: NCT00719849
Title: Transplantation of Unrelated Donor Umbilical Cord Blood in Patients With Hematological Malignancies Using a Non-Myeloablative Preparative Regimen
Brief Title: Donor Umbilical Cord Blood Transplant in Treating Patients With Advanced Hematological Cancer or Other Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: A new protocol was developed to replace this protocol in 2008, with removal of ATG and extension of MMF duration.
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Colleen Delaney, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012.00; FHCRC-2012.00 (Other: FHCRC Protocol Number); CDR0000597623 (Registry Identifier: PDQ); T32CA009515 (NIH)
Record Dates: First submitted 2008-07-19; First posted 2008-07-22 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases
Keywords: chronic myelogenous leukemia; acute lymphoblastic leukemia; acute myeloid leukemia; atypical chronic myeloid leukemia; chronic myelomonocytic leukemia; anaplastic large cell lymphoma; splenic marginal zone lymphoma; nodal marginal zone B-cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent childhood large cell lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; recurrent/refractory childhood Hodgkin lymphoma; childhood diffuse large cell lymphoma; childhood immunoblastic large cell lymphoma; refractory multiple myeloma; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; myelodysplastic/myeloproliferative disease; childhood myelodysplastic syndromes; recurrent childhood anaplastic large cell lymphoma; refractory anemia; refractory anemia with excess blasts; refractory anemia with ringed sideroblasts; refractory cytopenia with multilineage dysplasia; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage III childhood anaplastic large cell lymphoma; stage III childhood large cell lymphoma; stage IV childhood anaplastic large cell lymphoma; stage IV childhood large cell lymphoma; stage III adult Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; stage II multiple myeloma; stage III multiple myeloma; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV marginal zone lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; Waldenstrom macroglobulinemia; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; juvenile myelomonocytic leukemia; chronic eosinophilic leukemia; chronic idiopathic myelofibrosis; chronic neutrophilic leukemia; essential thrombocythemia; polycythemia vera
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Leukemia, Myelomonocytic, Chronic; Lymphoma, Large-Cell, Anaplastic; Lymphoma, B-Cell, Marginal Zone; Hodgkin Disease; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Dendritic Cell Sarcoma, Interdigitating; Mycosis Fungoides; Sezary Syndrome; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts; Waldenstrom Macroglobulinemia; Leukemia, Myelomonocytic, Juvenile; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Neutrophilic, Chronic; Thrombocythemia, Essential; Polycythemia Vera | interventions — Antilymphocyte Serum; Cyclophosphamide; Cyclosporine; fludarabine phosphate; Mycophenolic Acid; Cord Blood Stem Cell Transplantation; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cyclophosphamide/Fludarabine/TBI (Experimental): Subjects with hematological malignancies with prior autologous transplant, >2 cycles of multiagent chemotherapy, or severely immune suppressive therapy in last 3 months.
  Refractory leukemia and lymphoma in aplasia after induction chemotherapy or radioimmunoconjugated monoclonal antibody therapy.
  Interventions: Drug: cyclophosphamide; Drug: cyclosporine; Drug: fludarabine phosphate; Drug: mycophenolate mofetil; Procedure: umbilical cord blood transplantation; Radiation: total body irradiation
- Cyclophosphamide/Fludarabine/TBI/ATG (Experimental): Subjects with hematological malignancies with prior autologous transplant >12 mos or <1 cycle of multiagent chemotherapy or NO immune suppressive chemotherapy in last 3 months
  Interventions: Biological: anti-thymocyte globulin; Drug: cyclophosphamide; Drug: cyclosporine; Drug: fludarabine phosphate; Drug: mycophenolate mofetil; Procedure: umbilical cord blood transplantation; Radiation: total body irradiation

INTERVENTIONS:
Biological: anti-thymocyte globulin — 30mg/Kg Days -6 to -4
  Arms: Cyclophosphamide/Fludarabine/TBI/ATG
Drug: cyclophosphamide — 50 mg/Kg Day -6
Drug: cyclosporine — Patients will receive cyclosporine A (CSA) therapy beginning on Day -3 maintaining a trough level between 250 and 500 ng/mL. For adults the initial dose will be 2.5 mg/kg IV over 1 hour every 12 hours. For children < 40 kg the initial dose will be 2.5 mg/kg IV over 1 hour every 8 hours.
Drug: fludarabine phosphate — 40mg/m2 Days -6 to -2
Drug: mycophenolate mofetil — 1 gram every 8 hours for patients who are ≥ 40 kg. Pediatric patients (<40 kilograms) will receive MMF at the dose of 15 mg/kg/dose every 8 hours. Stop MMF at Day +30 or 7 days after engraftment, whichever day is later, if no acute GVHD.
Procedure: umbilical cord blood transplantation — Single or double unit umbilical cord blood transplant
Radiation: total body irradiation — 200 cGy Day -1

SUMMARY:
RATIONALE: Giving low doses of chemotherapy and total-body irradiation before a donor umbilical cord blood transplant helps stop the growth of cancer or abnormal cells. It may also stop the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving cyclosporine and mycophenolate mofetil before and after transplant may stop this from happening.

PURPOSE: This phase II trial is studying how well donor umbilical cord blood transplant with reduced intensity conditioning works in treating patients with advanced hematological cancer or other disease.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To estimate the probability of survival at 1 year in patients with advanced hematological malignancies or other diseases treated with non-myeloablative unrelated donor umbilical cord blood transplantation.

Secondary

* Six month non-relapse mortality.
* Chimerism at days 7, 14, 21, 28, 56, and 80, at 6 months, and at 1 and 2 years.
* To determine the incidence of neutrophil engraftment at day 42.
* To determine the incidence of platelet engraftment at 6 months.
* To determine the incidence of grade II-IV and III-IV acute graft-versus-host-disease (GVHD) at day 100.
* To determine the incidence of chronic GVHD at 1 year.
* To determine the incidence of clinically significant infections at 6 months and at 1 and 2 years.
* To determine the probability of progression-free survival at 1 and 2 years.
* To determine the probability of survival at 2 years.
* To determine the incidence of relapse or disease progression at 1 and 2 years.

OUTLINE: Patients are stratified according to disease status and prior therapy (hematologic malignancy or other disease that was treated with an autologous stem cell transplant or ≥ 2 courses of multiagent chemotherapy within the past 3 months vs hematologic malignancy or other disease that was treated with an autologous stem cell transplant > 12 months ago or with ≤ 1 course of multiagent chemotherapy or immunosuppressive chemotherapy within the past 3 months vs refractory leukemia or lymphoma for which patient was rendered aplastic either by induction chemotherapy or radioimmunoconjugated monoclonal antibody therapy).

* Conditioning regimen: Patients receive fludarabine phosphate IV over 1 hour on days -6 to -2 and cyclophosphamide IV on day -6. Patients also undergo total body irradiation on day -1. Some patients also receive anti-thymocyte globulin IV on days -6 to -4.
* Umbilical cord blood transplantation (UCBT): Patients undergo UCBT on day 0.
* Immunosuppressive therapy (graft-versus-host disease prophylaxis): Patients receive cyclosporine IV over 1 hour or orally (as tolerated) every 8 or 12 hours beginning on day -3 and continuing for approximately 6 months. Patients also receive mycophenolate mofetil IV every 8 hours on days -3 to 5 and then orally on days 6-30.

After completion of study treatment, patients are followed at 6 months and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of advanced hematologic malignancy or other disease not curable by conventional chemotherapy, including any of the following:

  * Acute myeloid leukemia in complete remission (CR)* (as defined by hematologic recovery, < 5% blasts in the bone marrow by morphology, and a cellularity of > 15%), meeting one of the following criteria:

    * In first complete remission (CR1) AND has high-risk disease as evidenced by any of the following:

      * Preceding myelodysplastic syndromes (MDS)
      * High-risk cytogenetics (e.g., monosomy 5 or 7, or as defined by referring institution treatment protocol)
      * Required > 2 courses of therapy to obtain CR
      * Erythroblastic or megakaryocytic leukemia
    * In second CR (CR2) or beyond
  * Acute lymphoblastic leukemia in CR* (as defined by hematologic recovery, < 5% blasts in the bone marrow by morphology, and a cellularity of > 15%), meeting one of the following criteria:

    * In CR1 AND has high-risk disease as evidenced by any of the following:

      * t(9;22), t(1;19), t(4;11), or other MLL rearrangements
      * Hyplodiploid
      * Required > 1 course of therapy to obtain CR
    * Beyond CR2
  * Chronic myelogenous leukemia (CML)

    * All types are allowed (except refractory blast crisis CML)
    * Patients in chronic phase CML must have failed or been intolerant to prior imatinib mesylate (Gleevec) or other tyrosine kinase inhibitors
  * MDS

    * Any subtype allowed (including refractory anemia [RA])
    * Severe pancytopenia or complex cytogenetics
    * Blasts must be < 5% (if blasts are ≥ 5%, pre-transplant induction therapy is required to reduce blast count to < 5%)
  * Large cell lymphoma, Hodgkin lymphoma, or multiple myeloma, meeting one of the following criteria:

    * Chemotherapy-sensitive disease that has failed prior therapy

      * Patients with large cell lymphoma or Hodgkin lymphoma must not have progressive disease during salvage therapy (stable disease allowed provided it is non-bulky)
    * Ineligible for an autologous stem cell transplant
  * Chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL), marginal zone B-cell lymphoma, or follicular lymphoma that has progressed after ≥ 2 prior therapies

    * Patients with bulky disease should be considered for debulking chemotherapy prior to transplant
    * Patients with refractory disease are eligible provided disease is non-bulky AND an estimated tumor doubling time is ≥ 1 month
  * Lymphoplasmacytic lymphoma, mantle cell lymphoma, or prolymphocytic leukemia

    * Chemotherapy-sensitive disease that was previously treated with initial therapy

      * Patients with mantle cell lymphoma must not have progressive disease during salvage therapy (stable disease allowed provided it is non-bulky)
  * Mycosis fungoides and Sezary syndrome
  * Bone marrow failure syndromes, except for Fanconi anemia
  * Myeloproliferative syndromes NOTE: *Patients for whom adequate marrow/biopsy specimens can not be obtained to determine remission status by morphologic assessment must have fulfilled criteria of remission (< 5% blasts by flow cytometry and recovery of peripheral blood counts with no circulating blasts)
* Ineligible for autologous stem cell transplant due to any of the following:

  * Prior autologous stem cell transplant
  * Inadequate autologous stem cell harvest
  * Inability to withstand a myeloablative preparative regimen
  * Clinically aggressive/high-risk disease
* No evidence of progressive disease by imaging modalities or biopsy (persistent PET scan activity allowed provided there are no CT scan changes indicating progression)
* Acute leukemia that is refractory, persistent, or relapsed (defined as > 5% blasts in normocellular bone marrow) allowed provided patient was rendered aplastic either by induction chemotherapy or radioimmunoconjugated monoclonal antibody therapy
* Patients with stable disease are eligible provided the largest residual nodal mass is approximately < 5 cm (largest residual mass must represent a 50% reduction and be approximately < 7.5 cm for patients who have responded to prior therapy)
* No active CNS malignancy
* Umbilical cord blood (UCB) donor available

  * UCB graft matched at 4/6 HLA-A, -B, and -DRB1 antigens with the recipient

    * May include 0-2 antigen mismatches at the A, B, or DRB1 loci
    * Unit selection based on cryopreserved nucleated cell dose and HLA-A, -B, and -DRB1 using intermediate resolution A, B antigen and DRB1 allele typing
  * If 2 UCB units are required to reach the target cell dose, each unit must be a 3/6 HLA-A, -B, and -DRB1 antigen match to each other, as well as a 4/6 antigen match to the recipient
  * No 5-6/6 HLA-A, -B, and -DRB1 matched sibling donor available

PATIENT CHARACTERISTICS:

* Karnofsky performance status (PS) 60-100% OR Lansky PS 50-100%
* Creatinine ≤ 2.0 mg/dL (adults) OR creatinine clearance > 40 mL/min (pediatrics)

  * Adult patients with a creatinine > 1.2 mg/dL or a history of renal dysfunction must have an estimated creatinine clearance of > 40 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* LVEF ≥ 35%
* DLCO > 30% predicted
* No requirement for O_2
* No decompensated congestive heart failure
* No uncontrolled arrhythmia
* None of the following liver diseases or conditions:

  * Fulminant liver failure
  * Cirrhosis with evidence of portal hypertension or bridging fibrosis
  * Alcoholic hepatitis
  * Esophageal varices
  * History of bleeding esophageal varices, hepatic encephalopathy, or correctable hepatic synthetic dysfunction as evidenced by prolongation of the prothrombin time
  * Ascites related to portal hypertension
  * Bacterial or fungal abscess
  * Biliary obstruction
  * Chronic viral hepatitis with total serum bilirubin > 3 mg/dL
  * Symptomatic biliary disease
* Recent mold infection (e.g., Aspergillus) allowed provided patient received ≥ 30 days of appropriate treatment AND infection is controlled and cleared by Infectious Disease
* No evidence of HIV infection or known HIV-positive serology
* No uncontrolled viral or bacterial infection

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 3 months since prior myeloablative stem cell transplantation

Max Age: 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2005-11; Primary Completion 2008-11 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Delaney, MD, MSC, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cyclophosphamide/Fludarabine/TBI: Subjects with hematological malignancies with prior autologous transplant, >2 cycles of multiagent chemotherapy, or severely immune suppressive therapy in last 3 months, OR patients with refractory leukemia and lymphoma in aplasia after induction chemotherapy or radioimmunoconjugated monoclonal antibody therapy.
  * Cyclophosphamide 50 mg/Kg Day -6
  * Fludarabine 40mg/m2 Days -6 to -2
  * TBI 200 cGy Day -1
  Immune suppression begin Day -3: cyclosporine and mycophenolate mofetil
- Cyclophosphamide/Fludarabine/TBI/ATG: Subjects with hematological malignancies with prior autologous transplant >12 mos or <1 cycle of multiagent chemotherapy or NO immune suppressive chemotherapy in last 3 months, and who should receive ATG as part of their conditioning regimen.
  * Cyclophosphamide 50 mg/Kg Day -6
  * Fludarabine 40mg/m2 Days -6 to -2
  * TBI 200 cGy Day -1
  * Equine ATG 30mg/Kg Days -6 to -4
  Immune suppression begin Day -3: cyclosporine and mycophenolate mofetil
Period: Overall Study
Arm/Group | Cyclophosphamide/Fludarabine/TBI | Cyclophosphamide/Fludarabine/TBI/ATG
Started | 4 | 9
Completed | 4 | 8
Not Completed | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cyclophosphamide/Fludarabine/TBI | Cyclophosphamide/Fludarabine/TBI/ATG | Total
Number analyzed (Participants) | 4 | 9 | 13
Age, Continuous [Mean (Full Range); unit: years] | 52.5 [24 to 67] | 55.1 [37 to 68] | 53.6 [24 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 3 | 5 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 4 | 7 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 9 | 13
Disease Diagnosis [Count of Participants; unit: Participants]
  AML (Acute Myeloid Leukemia) | 4 | 5 | 9
  CML (Chronic Myeloid Leukemia) | 0 | 1 | 1
  NHL (Non-Hodgkin's Lymphoma) | 0 | 1 | 1
  MDS (Myelodysplastic Syndromes) | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Probability of Survival at 1 Year
Description: Kaplan-Meier estimate of the probability of survival at 1 year
Time Frame: 1 year post transplant
Measure: Number (95% Confidence Interval); unit: survival probability
Groups:
- Cyclophosphamide/Fludarabine/TBI: Subjects with hematological malignancies with prior autologous transplant, >2 cycles of multiagent chemotherapy, or severely immune suppressive therapy in last 3 months, OR subjects with refractory leukemia and lymphoma in aplasia after induction chemotherapy or radioimmunoconjugated monoclonal antibody therapy.
  * Cyclophosphamide 50 mg/Kg Day -6
  * Fludarabine 40mg/m2 Days -6 to -2
  * TBI 200 cGy Day -1
  Immune suppression: begin Day -3 cyclosporine and mycophenolate mofetil
- Cyclophosphamide/Fludarabine/TBI/ATG: Subjects with hematological malignancies with prior autologous transplant >12 mos or <1 cycle of multiagent chemotherapy or NO immune suppressive chemotherapy in last 3 months.
  * Cyclophosphamide 50 mg/Kg Day -6
  * Fludarabine 40mg/m2 Days -6 to -2
  * TBI 200 cGy Day -1
  * Equine ATG 30mg/Kg Days -6 to -4
  Immune suppression: begin Day -3 cyclosporine and mycophenolate mofetil
Arm/Group | Cyclophosphamide/Fludarabine/TBI | Cyclophosphamide/Fludarabine/TBI/ATG
Number analyzed (Participants) | 4 | 8
survival probability | 0.25 [0.046 to 1.000] | 0.50 [0.25 to 1.00]

2. Secondary Outcome: Probability of Survival at 2 Years
Description: Kaplan-Meier estimate of the probability of survival at 2 years
Time Frame: 2 years post transplant
Measure: Number (95% Confidence Interval); unit: survival probability
Arm/Group | Cyclophosphamide/Fludarabine/TBI | Cyclophosphamide/Fludarabine/TBI/ATG
Number analyzed (Participants) | 4 | 8
survival probability | 0.25 [0.046 to 1.000] | 0.38 [0.15 to 0.92]

3. Secondary Outcome: Incidence of Non-relapse Mortality at 6 Months
Description: Number of Participants with Non-relapse Mortality at 6 Months
Time Frame: 6 months post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Cyclophosphamide/Fludarabine/TBI | Cyclophosphamide/Fludarabine/TBI/ATG
Number analyzed (Participants) | 4 | 8
Participants | 2 | 2

4. Secondary Outcome: Chimerism
Description: Count of participants who experienced dominance of one cord blood unit (defined by >or= 95% contribution of one cord blood unit to BM and all PB fractions -- CD3+, CD33+, CD56+, and CD19+) at 7 days, 14 days, 21 days, 28 days, 56 days, and 80 days, 6 months, 1 and 2 years post transplant.
Time Frame: 7 days, 14 days, 21 days, 28 days, 56 days, and 80 days, 6 months, 1 and 2 years post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Cyclophosphamide/Fludarabine/TBI | Cyclophosphamide/Fludarabine/TBI/ATG
Number analyzed (Participants) | 4 | 8
Participants
  Day 7 | 0 | 0
  Day 14 | 0 | 0
  Day 21 | 1 | 1
  Day 28 | 1 | 5
  Day 56 | 1 | 5
  Day 80 | 1 | 6
  6 months | 2 | 7
  1 year | 2 | 7
  2 years | 2 | 7

5. Secondary Outcome: Incidence of Neutrophil Engraftment at Day 42
Description: Number of participants with neutrophil engraftment at day 42
Time Frame: Day 42 post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Cyclophosphamide/Fludarabine/TBI | Cyclophosphamide/Fludarabine/TBI/ATG
Number analyzed (Participants) | 4 | 8
Participants | 3 | 7

6. Secondary Outcome: Incidence of Platelet Engraftment at 6 Months
Description: Number of participants with platelet engraftment at 6 months
Time Frame: 6 months post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Cyclophosphamide/Fludarabine/TBI | Cyclophosphamide/Fludarabine/TBI/ATG
Number analyzed (Participants) | 4 | 8
Participants | 2 | 2

7. Secondary Outcome: Incidence of Grade II-IV Acute Graft-versus-host-disease (GVHD) at Day 100
Description: Number of participants with Grade II-IV acute graft-versus-host-disease (GVHD) at day 100.
  Acute GVHD Staging and Grading:
  Overall grade 1: stage 1-2 skin, no liver or gut Overall grade 2: stage 3 skin or stage 1 liver or stage 1 gut Overall grade 3: stage 4 skin or stage 2-4 liver or stage 2-4 gut (without GVHD as a major contributing cause of death) Overall grade 4: stage 4 skin or stage 2-4 liver or stage 2-3 gut (with GVHD as a major contributing cause of death)
Time Frame: Day 100 post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Cyclophosphamide/Fludarabine/TBI | Cyclophosphamide/Fludarabine/TBI/ATG
Number analyzed (Participants) | 4 | 8
Participants | 3 | 6

8. Secondary Outcome: Incidence of Grade III-IV Acute Graft-versus-host-disease (GVHD) at Day 100
Description: Number of participants with Grade III-IV acute graft-versus-host-disease (GVHD) at day 100.
  Acute GVHD Staging and Grading:
  Overall grade 1: stage 1-2 skin, no liver or gut Overall grade 2: stage 3 skin or stage 1 liver or stage 1 gut Overall grade 3: stage 4 skin or stage 2-4 liver or stage 2-4 gut (without GVHD as a major contributing cause of death) Overall grade 4: stage 4 skin or stage 2-4 liver or stage 2-3 gut (with GVHD as a major contributing cause of death)
Time Frame: Day 100 post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Cyclophosphamide/Fludarabine/TBI | Cyclophosphamide/Fludarabine/TBI/ATG
Number analyzed (Participants) | 4 | 8
Participants | 2 | 1

9. Secondary Outcome: Incidence of Chronic Graft-versus-host-disease (GVHD) at 1 Year
Description: Number of participants with chronic graft-versus-host-disease (GVHD) at 1 year.
  Clinical Limited cGVHD
  1. Oral abnormalities consistent with cGVHD, a positive skin or lip biopsy, and no other manifestations of cGVHD.
  2. Mild liver test abnormalities (alkaline phosphatase <2 x upper limit of normal, AST or ALT <3 x upper limit of normal and total bilirubin <1.6) with positive skin or lip biopsy, and no other manifestations of cGVHD.
  3. Less than 6 papulosquamous plaques, macular-papular or lichenoid rash involving <20% of body surface area (BSA), dyspigmentation involving <20% BSA, or erythema involving <50% BSA, positive skin biopsy, and no other manifestations of cGVHD.
  4. Ocular sicca (Schirmer's test <5mm with no more than minimal ocular symptoms), positive skin or lip biopsy, and no other manifestations of cGVHD.
  5. Vaginal or vulvar abnormalities with positive biopsy, and no other manifestations of cGVHD.
Time Frame: 1 year post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Cyclophosphamide/Fludarabine/TBI | Cyclophosphamide/Fludarabine/TBI/ATG
Number analyzed (Participants) | 4 | 8
Participants | 0 | 3

10. Secondary Outcome: Incidence of Clinically Significant Infections at 6 Months
Description: Number of participants with clinically significant infections at 6 months
Time Frame: 6 months post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Cyclophosphamide/Fludarabine/TBI | Cyclophosphamide/Fludarabine/TBI/ATG
Number analyzed (Participants) | 4 | 8
Participants | 3 | 3

11. Secondary Outcome: Incidence of Clinically Significant Infections at 1 Year
Description: Number of participants with clinically significant infections at 1 year
Time Frame: 1 year post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Cyclophosphamide/Fludarabine/TBI | Cyclophosphamide/Fludarabine/TBI/ATG
Number analyzed (Participants) | 4 | 8
Participants | 3 | 3

12. Secondary Outcome: Incidence of Clinically Significant Infections at 2 Years
Description: Number of participants with clinically significant infections at 2 years
Time Frame: 2 years post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Cyclophosphamide/Fludarabine/TBI | Cyclophosphamide/Fludarabine/TBI/ATG
Number analyzed (Participants) | 4 | 8
Participants | 3 | 3

13. Secondary Outcome: Probability of Progression-free Survival at 1 Year
Description: Kaplan-Meier estimate of the probability of progression-free survival at 1 year
Time Frame: 1 year post transplant
Measure: Number (95% Confidence Interval); unit: progression free survival probability
Arm/Group | Cyclophosphamide/Fludarabine/TBI | Cyclophosphamide/Fludarabine/TBI/ATG
Number analyzed (Participants) | 4 | 8
progression free survival probability | 0.25 [0.046 to 1.000] | 0.38 [0.15 to 0.92]

14. Secondary Outcome: Probability of Progression-free Survival at 2 Years
Description: Kaplan-Meier estimate of the probability of progression-free survival at 2 years
Time Frame: 2 years post transplant
Measure: Number (95% Confidence Interval); unit: progression free survival probability
Arm/Group | Cyclophosphamide/Fludarabine/TBI | Cyclophosphamide/Fludarabine/TBI/ATG
Number analyzed (Participants) | 4 | 9
progression free survival probability | 0.25 [0.046 to 1.000] | 0.25 [0.075 to 0.83]

15. Secondary Outcome: Incidence of Relapse at 1 Year
Description: Number of participants with relapse at 1 year.
  Patients with leukemia and lymphoma involving the BM and multiple myeloma will have this done by BM biopsy and additional special studies such as cytogenetics or flow cytometry as appropriate. Patients with lymphoma and myeloma will have radiology studies such as plain X-rays or CT scans and/or other studies such as blood tumor markers to document presence or absence of disease as clinically indicated.
Time Frame: 1 year post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Cyclophosphamide/Fludarabine/TBI | Cyclophosphamide/Fludarabine/TBI/ATG
Number analyzed (Participants) | 4 | 8
Participants | 1 | 4

16. Secondary Outcome: Incidence of Relapse at 2 Years
Description: Number of participants with relapse at 2 years.
  Patients with leukemia and lymphoma involving the BM and multiple myeloma will have this done by BM biopsy and additional special studies such as cytogenetics or flow cytometry as appropriate. Patients with lymphoma and myeloma will have radiology studies such as plain X-rays or CT scans and/or other studies such as blood tumor markers to document presence or absence of disease as clinically indicated.
Time Frame: 2 years post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Cyclophosphamide/Fludarabine/TBI | Cyclophosphamide/Fludarabine/TBI/ATG
Number analyzed (Participants) | 4 | 8
Participants | 1 | 5

ADVERSE EVENTS:
Arm/Group | Cyclophosphamide/Fludarabine/TBI | Cyclophosphamide/Fludarabine/TBI/ATG
Serious Adverse Events (participants affected / at risk) | 3/4 | 8/9
Other Adverse Events (participants affected / at risk) | 2/4 | 3/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cyclophosphamide/Fludarabine/TBI (N=4) | Cyclophosphamide/Fludarabine/TBI/ATG (N=9)
Death (Investigations) | 3 (3) | 8 (8)
Relapse of underlying disease (Blood and lymphatic system disorders) | 1 (1) | 5 (5)
Congestive heart failure (Cardiac disorders) | 1 (1) | 0 (0)
MSOF leading to death (General disorders) | 1 (1) | 0 (0)
Fever of unknown etiology (General disorders) | 1 (1) | 3 (3)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Creatinine Phosphokinase (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Infection with grade 3 ANC - blood (Infections and infestations) | 1 (1) | 0 (0)
Infection with grade 3 ANC - lungs (Infections and infestations) | 1 (1) | 0 (0)
ARDS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Infection with normal ANC - blood (Infections and infestations) | 0 (0) | 1 (1)
Opportunistic infection associated with lymphopenia (Infections and infestations) | 0 (0) | 1 (1)
Obstruction, GI - biliary tree (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 2 (4)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1)
Failure to engraft by day 42 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Encephalitis HHV6 (Infections and infestations) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Secondary graft failure (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Pulmonary VOD (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cyclophosphamide/Fludarabine/TBI (N=4) | Cyclophosphamide/Fludarabine/TBI/ATG (N=9)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Glucose, serum-high (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Potassium, serum-high (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Potassium, serum-low (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Sodium, serum-low (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Platelets (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Thrombus (Vascular disorders) | 0 (0) | 1 (1)
Phosphate, serum-low (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Magnesium, serum-high (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutrophils (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Leukocytes (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Infection with grade 2 ANC - skin (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC - blood (Infections and infestations) | 0 (0) | 1 (1)
Infection with grade 4 ANC - blood (Infections and infestations) | 0 (0) | 1 (1)
Infection with grade 4 ANC - oral (Infections and infestations) | 0 (0) | 1 (1)
AST (Metabolism and nutrition disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No